CLINICAL TRIAL: NCT04656782
Title: Towards Standardization of mCRC Imaging - an EORTC-endorsed, Prospective European Multicenter Imaging Survey and Imaging Protocol
Brief Title: EORTC-endorsed, Prospective European Multicenter Imaging Survey and Protocol
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: EORTC Imaging Group (Unknown); EORTC Gastrointestinal Tract Cancer Cooperative Group (Other); European Society of Oncologic Imaging (ESOI) (Unknown); European Society of Gastrointestinal and Abdominal Radiology (ESGAR) (Unknown)
Responsible Party: Principal Investigator, Marcus Unterrainer, Resident, Department of Radiology, University Hospital, LMU Munich, Ludwig-Maximilians - University of Munich
Other Study IDs: EORTC imaging survey
Record Dates: First submitted 2020-11-25; First posted 2020-12-07 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Computed Tomography (CT); Radiomics; Delphi Survey; PET/CT; Expert Panelists; Standardization; Imaging protocol
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expert panelists: Expert panelists will be recruited from EORTC Imaging Group, EORTC GI Group, ESOI and ESGAR and will actively participate in the imaging survey rounds.
  Interventions: Other: Imaging survey
- Facilitators: The two central facilitators will moderate and guide the survey rounds. Blinded results will be forwarded to the expert panelists by the facilitators. Further Survey rounds will be adapted by the facilitators according to the previous answers given by the panelists.
  Interventions: Other: Facilitation

INTERVENTIONS:
Other: Imaging survey — Participation as expert panelist in the imaging survey.
  Groups: Expert panelists
Other: Facilitation — Moderation and evaluation of the expert panel's answers. Adoption and moderation of further survey rounds.
  Groups: Facilitators

SUMMARY:
A prospective, multicenter imaging Delphi survey among European radiological societies for mCRC imaging standardization.

DETAILED DESCRIPTION:
BACKGROUND: Computed Tomography (CT) is the imaging reference standard for initial staging and response assessment in randomized, controlled clinical trials (RCT) dealing with metastatic colorectal cancer (mCRC). However, comparability of imaging data among recruiting centers in RCTs is highly hampered by diverging imaging protocols and different technical specifications. Over the last years, analysis of radiomic features in mCRC patients has gained increasing interest for image evaluation beyond the mere assessment of extent. Also, these radiomic features are highly susceptible to technical parameters such as slice thickness. Hence, comparability of radiomic features among recruiting centers are also highly limited due to diverging imaging protocols.

AIMS: This prospective, multicenter imaging survey aims at assessing current differences regarding mCRC CT imaging protocols and technical specifications among large academic sites in Europe and at drafting a consensus imaging protocol endorsed by the European Organisation for Research and Treatment of Cancer (EORTC).

METHODS: This survey will be in close cooperation of the EORTC Imaging Group, EORTC Gastro-intestinal Tract Group, European Society of Oncologic Imaging (ESOI) and European Society of Gastrointestinal and Abdominal Radiology (ESGAR). Among the EORTC Imaging Group, EORTC Gastro-intestinal Tract Group, ESOI and ESGAR, imaging experts will be prospectively recruited and will serve as expert panelists in this prospective survey. Following the Delphi approach for survey conduction, several survey rounds will be performed. The answers of each survey round will be analyzed by the survey facilitators, blinded results will then be forwarded to the expert panelists prior to every following survey round. Statements / answers can then be modified by the expert panelists in the following survey round.

ELIGIBILITY:
Inclusion Criteria:

* Researchers / academics with expertise in gastro-intestinal / oncologic imaging
* Association with EORTC Imaging Group, EORTC GI Group, ESGAR or ESOI.

Exclusion Criteria:

* Participants not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Imaging experts will serve as expert panelists in the Delphi Survey and will undergo several rounds of blinded questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-01-26 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized imaging protocol consensus among panelists | 6 months after finalization of the last survey round
  Standardized imaging protocol among panelists after multiple rounds of Delphi consensus survey (technical parameters, e. g. contrast phases, oral contrast etc.)

SECONDARY OUTCOMES:
Description of technical comparability of datasets for radiomic and AI analyses | 6 months after finalization of the last survey round
  During the Delphi-survey, local information regarding technical specifications in their departments (e. g. vendor, scanner type, contrast phases, slice thickness, oral contrast, kV, etc.) will be enquired. The results will be reported as descriptive statistics, e. g. on percentage distribution of a particular technical feature. This analyses will be performed with special regards to technical parameters that knowingly have a major impact on reproducibility of Radiomics features.
Description of heterogeneity of mCRC imaging protocols | 6 months after finalization of the last survey round
  During the Delphi-survey, local information regarding technical specifications in their departments (e. g. vendor, scanner type, contrast phases, slice thickness, oral contrast, kV, etc.) will be enquired. The results will be reported as descriptive statistics, e. g. on percentage distribution of a particular technical feature.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Unterrainer, Principal Investigator — Dept. of Radiology, University Hospital, LMU Munich; Wolfgang G Kunz, Principal Investigator — Dept. of Radiology, University Hospital, LMU Munich
Locations (1):
- Dept. of Radiology, University Hospital, LMU Munich, Munich, Bavaria, Germany

REFERENCES:
- See also: EORTC Imaging Group — https://www.eortc.org/blog/category/imaging-group/
- See also: EORTC Gastrointestinal Tract Cancer Group — https://www.eortc.org/blog/category/gastrointestinal-tract-cancer-group/
- See also: European Society of Oncologic Imaging — http://www.esoi-society.org/
- See also: European Society of Gastrointestinal and Abdominal Radiology — https://www.esgar.org/